CLINICAL TRIAL: NCT01553136
Title: 1/2-Multi-site Study: Varenicline Treatment of Alcohol Dependent Smokers
Brief Title: Varenicline Treatment of Alcohol Dependence in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Columbia University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1106008598; 1R01AA020388-01A1 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-03-13 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2018-10

CONDITIONS: Alcoholism; Alcohol Abuse; Smoking; Alcohol Drinking
Keywords: alcohol-related disorders; Cholinergic Drugs; varenicline; Chantix
MeSH Terms: conditions — Alcoholism; Smoking; Alcohol Drinking; Alcohol-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Varenicline
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — 0.5 mg once per day for Days 1 to 3, 0.5 mg twice per day for Days 4 to 7, then two 0.5 mg tablets (1 mg) twice per day
  Other Names: Chantix

SUMMARY:
The purpose of this study is to determine whether varenicline is effective in the treatment of alcohol dependence in smokers.

DETAILED DESCRIPTION:
Building upon knowledge about the role of nicotinic acetylcholine receptors in alcohol drinking and smoking, varenicline, a smoking cessation treatment that targets these receptors, will be tested as a potential treatment for alcohol dependent smokers seeking alcohol treatment.

ELIGIBILITY:
Inclusion Criteria:

* are 18 - 70 years of age and seeking treatment of alcohol drinking;
* meet DSM-IV TR Criteria for Alcohol Dependence
* report smoking 100 cigarettes or more in their lifetime and currently smoke at least twice weekly on average in the past 90 days and have a urinary cotinine level of > 30ng/mL by semi-quantitative urinalysis or equivalent plasma cotinine level (> 6 ng/mL);
* report heavy drinking on at least 2 days on average per week (i.e., ≥ 4 drinks on an occasion for women and ≥ 5 drinks for men) for the past 90 days and no more than 7 consecutive days of abstinence at intake.

Exclusion Criteria:

* exhibit current, clinically significant physical disease or abnormality based on medical history, physical examination, or routine laboratory evaluation including:

  * any unexplained elevations in liver enzymes (i.e., transaminases, bilirubin)
  * clinically significant, unstable cardiovascular disease/uncontrolled hypertension
  * hepatic or renal impairment
  * severe obstructive pulmonary disease
  * diabetes mellitus requiring insulin or certain oral medications (i.e., sulfonylureas) and an A1C hemoglobin test score of > 7 for participants not prescribed these medications
  * baseline systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 95 mm Hg
* have a history of cancer (except treated basal cell or squamous cell carcinoma of the skin)
* have a history of serious hypersensitivity reactions or skin reactions to varenicline;
* exhibit serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality disorder, organic mood or mental disorders by history or psychological examination
* report current suicidal ideation (past 6 months) or lifetime hx of suicidal behavior assessed with the Columbia Suicide Severity Rating Scale 60; or risk for aggression using a cut-off of 15 or more on the Overt Aggression Scale - Modified Aggression Scale or 6 or more on the OAS-M Irritability Subscale 61.
* have used any psychotropic drug in the past month, except individuals who are on a stable dose of a Selective Serotonin Reuptake Inhibitor for at least two months or who report occasional use of prescription sleep aids that they are willing to discontinue;
* have a current DSM-IV diagnosis of drug dependence other than nicotine or alcohol
* are at risk for an alcohol withdrawal syndrome as evidenced by:

  * a history of seizures, delirium, or hallucinations during alcohol withdrawal
  * a Clinical Institute Withdrawal Assessment scale 62 score of > 8,
  * report drinking to avoid withdrawal symptoms
  * have required medical treatment of alcohol withdrawal within the past 6 months
* have used another investigational drug within 30 days or have used medications to treat alcohol (e.g., naltrexone, topiramate, acamprosate, disulfiram) or nicotine use (e.g., clonidine, varenicline, bupropion, nicotine replacement) in the past 3 months or intend to use these medications;prior use of nicotine replacement in situations where smoking is not permitted (e.g., planes) without the intention to quit smoking is not exclusionary;
* intend to donate blood or blood products during the treatment phase of the study
* have a Body Mass Index (calculated as weight in kilograms divided by the square of height in meters) less than 15 or greater than 39.99 or weight less than 45 kg;
* are a female of childbearing potential who is pregnant, nursing, or not practicing effective contraception (oral, injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, PhD, Principal Investigator — Yale University; Allen Zweben, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center - Substance Abuse Treatment Unit, New Haven, Connecticut
  - Parallax Center, New York, New York

REFERENCES:
- [Derived] Bold KW, Zweben A, Fucito LM, Piepmeier ME, Muvvala S, Wu R, Gueorguieva R, O'Malley SS. Longitudinal Findings from a Randomized Clinical Trial of Varenicline for Alcohol Use Disorder with Comorbid Cigarette Smoking. Alcohol Clin Exp Res. 2019 May;43(5):937-944. doi: 10.1111/acer.13994. Epub 2019 Mar 21. PMID 30817018
- [Derived] O'Malley SS, Zweben A, Fucito LM, Wu R, Piepmeier ME, Ockert DM, Bold KW, Petrakis I, Muvvala S, Jatlow P, Gueorguieva R. Effect of Varenicline Combined With Medical Management on Alcohol Use Disorder With Comorbid Cigarette Smoking: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):129-138. doi: 10.1001/jamapsychiatry.2017.3544. PMID 29261824

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Sugar Pill
Started | 64 | 67
Completed Treatment (These data reflect those that had complete alcohol timeline data.) | 55 | 52
Completed (The completed participants reflect those that continued on medication.) | 48 | 45
Not Completed | 16 | 22
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 4 | 10
Not completed — Physician Decision | 2 | 3
Not completed — Scheduling Difficulties | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Varenicline | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.7) | 43.6 (11.7) | 42.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 47 | 45 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 57 | 59 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Multiple races ("Other") are reported in the 'More than 1 Race' row.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 35 | 34 | 69
    White | 24 | 26 | 50
    More than one race | 8 | 4 | 12
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days During the Last 8 Weeks of Treatment
Description: The percentage of days of heavy drinking will be examined over the final 8 weeks of the study averaged by month (weeks 9-12 and weeks 13-16). A heavy drinking day is defined as 5 or more standard drinks for men and 4 or more standard drinks for women. A standard drink contains approximately 0.6 fluid ounces of pure alcohol.
Time Frame: weeks 9-12
Measure: Mean (Standard Error); unit: log transformed percentage of days
Groups:
- Placebo: Placebo: once per day for Days 1 to 3, twice per day for the remaining days
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 64 | 67
log transformed percentage of days | 2.07 (0.23) | 2.25 (0.20)

2. Primary Outcome: Percentage of Heavy Drinking Days During the Last 8 Weeks of Treatment
Description: as for outcome 1
Time Frame: weeks 13-16
Measure: Mean (Standard Error); unit: log transformed percentage of days
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 64 | 67
log transformed percentage of days | 1.99 (0.22) | 2.09 (0.21)

3. Primary Outcome: Percentage of Heavy Drinking Days During the Last 8 Weeks of Treatment
Description: The percentage of days of heavy drinking will be examined over the final 8 weeks of the study. A heavy drinking day is defined as 5 or more standard drinks for men and 4 or more standard drinks for women. A standard drink contains approximately 0.6 fluid ounces of pure alcohol. Presented here is the average of the 8 weeks (reported as week 17 originally).
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 64 | 67
percentage of heavy drinking days | 2.40 (0.21) | 2.28 (0.21)

4. Secondary Outcome: Smoking Abstinence
Description: Smoking abstinence is defined by self-reported abstinence from smoking for the last four weeks of treatment (weeks 13-16) and a urine cotinine level less than 15ng/mL measured at week 17.
Time Frame: Weeks 13-16
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 64 | 67
Participants | 8 | 0

5. Secondary Outcome: Drinking Related Consequences
Description: A self-report measure of negative consequences from drinking will be administered and the total score are analyzed. The ImBIBe, a measure of alcohol consequences based on the Drinker Inventory of Consequences (DRINC) was used. The DRINC total score has a range from 0-45, 45 being the highest score (or greatest number of negative consequences).
Time Frame: End of treatment (Week 17)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 64 | 67
units on a scale | 1.29 (0.03) | 1.40 (0.03)

ADVERSE EVENTS:
Arm/Group | Varenicline | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/67
Serious Adverse Events (participants affected / at risk) | 2/64 | 0/67
Other Adverse Events (participants affected / at risk) | 47/64 | 46/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=64) | Sugar Pill (N=67)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Behavior (Psychiatric disorders) | 1 (1) | 0 (0) — Patient was admitted to alcohol rehabilitation after trying to 'dink self to death'.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=64) | Sugar Pill (N=67)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Anxiety (Psychiatric disorders) | 8 | 6
Depression (Psychiatric disorders) | 11 | 8
Disturbance in Attention (Nervous system disorders) | 6 | 5
Fatigue (Nervous system disorders) | 9 | 13
Headache (Nervous system disorders) | 16 | 15
Insomnia (Nervous system disorders) | 10 | 9
Irritability (Nervous system disorders) | 20 | 20
Abnormal Dreams (Nervous system disorders) | 28 | 15
Rhinorrhea (Ear and labyrinth disorders) | 11 | 9
Acid Reflux (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 4 | 9
Decreased Appetite (Gastrointestinal disorders) | 11 | 11
Diarrhea (Gastrointestinal disorders) | 4 | 10
Dry Mouth (Gastrointestinal disorders) | 10 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Flatulence (Gastrointestinal disorders) | 10 | 8
Taste Perversion (Gastrointestinal disorders) | 3 | 5
Increased Appetite (Gastrointestinal disorders) | 11 | 10
Increased Bowel Movements (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 25 | 18
Vomiting (Gastrointestinal disorders) | 4 | 7
Frequent Urination (Renal and urinary disorders) | 12 | 7
Joint Pain and Swelling (Musculoskeletal and connective tissue disorders) | 3 | 5
Blurred Vision (Eye disorders) | 4 | 2
Diaphoresis (General disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes